CLINICAL TRIAL: NCT03560505
Title: A Prospective Study of High-resolution Ultrasonography in Examination of Lower Extremity Peripheral Nerves in Patients With Compression Neuropathies and in Healthy Controls.
Brief Title: High-resolution Ultrasound in Lower Extremity Nerves and Common Fibular Neuropathies.
Status: Completed | Type: Observational
Sponsor: Sándor Beniczky (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: USCF
Record Dates: First submitted 2018-06-07; First posted 2018-06-18 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2018-06

CONDITIONS: Ultrasonography; Peroneal Neuropathies
Keywords: Ultrasound reference material; Sensitivity; Specificity; Common fibular compression neuropathy; Type 2 diabetes polyneuropathy; Intra-rater reliability; Inter-rater reliability
MeSH Terms: conditions — Peroneal Neuropathies; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Common fibular compression neuropathy: Patients referred for electrophysiological assessment of common fibular compression neuropathy with subsequent confirmation of referral diagnosis.
  Intervention: Ultrasound protocol.
  Interventions: Diagnostic Test: Ultrasound protocol
- Type 2 diabetes polyneuropathy: Patients with type 2 diabetes referred for polyneuropathy involving the common fibular nerve with subsequent confirmation of referral diagnosis.
  Intervention: Ultrasound protocol.
  Interventions: Diagnostic Test: Ultrasound protocol

INTERVENTIONS:
Diagnostic Test: Ultrasound protocol — High-resolution ultrasound protocol at pre-defined sites bilaterally. Pre-defined sites: Sciatic nerve (proximal and distal), tibial nerve (proximal and distal), common fibular nerve (proximal and distal), superficial fibular nerve (proximal and distal) and sural nerve (proximal and distal).

SUMMARY:
This study establishes reference material of selected lower extremity nerves at pre-defined sites with high-resolution ultrasound. Furthermore in this study, high-resolution ultrasound of patients with common fibular compression neuropathy and patients with type 2 diabetic polyneuropathy involving the common fibular nerve will be examined and compared to healthy controls. High-resolution ultrasound measurements will be correlated with history, clinical information and electrophysiological data.

DETAILED DESCRIPTION:
The usual diagnostic work-up of patients referred for lower-extremity neuropathy includes clinical examination, biochemical tests (blood and cerebrospinal fluid), electrophysiological assessment and if necessary nerve biopsy. The electrophysiological assessment usually consists of nerve conduction studies (NCS) and electromyography (EMG). While electrophysiological measurements generally give information about the function of nerves, high-resolution ultrasound may provide information about the structure of nerves.

High-resolution ultrasound examination has shown promising results as a supplementary tool in the diagnostic work-up of various peripheral neuropathies. The clinical utility of ultrasound in the diagnosis of common fibular neuropathies, however, calls for further elucidation.

This study establishes reference material of selected lower extremity nerves at pre-defined sites with high-resolution ultrasound. Furthermore in this study, high-resolution ultrasound of patients with common fibular compression neuropathy and patients with type 2 diabetic polyneuropathy involving the common fibular nerve will be examined and compared to healthy controls, as well as each other. High-resolution ultrasound measurements will be correlated with history, clinical information and electrophysiological data.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes polyneuropathy common fibular nerve affection or
* Common fibular nerve compression neuropathy

Exclusion Criteria:

* Lumbar radiculopathy
* Other competing lower extremity peripheral neuropathy
* Peripheral vascular disease
* Hypothyroidism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with common fibular compression neuropathy and patients with type 2 diabetes polyneuropathy involving the common fibular nerve
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Nerve cross-sectional area (CSA) | 1 year
  The nerve cross-sectional area within the hyperechoic epineurium measured with ultrasound machine software.
Common fibular nerve fascicle properties | 1 year
  The amount of visible fascicles and fascicle CSA of the common fibular nerve at measurement sites.

CONTACTS AND LOCATIONS:
Overall Officials: Erisela Qerama Montvilas, MD, PhD, Study Director — Department of Clinical Neurophysiology, Aarhus University Hospital
Locations (1):
- Department of Clinical Neurophysiolgy, Department of Neurology, Aarhus University Hospital, Aarhus, Denmark